CLINICAL TRIAL: NCT01805713
Title: Biomarkers of Injury and Destruction in the Cystic Fibrosis Lung
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Minnesota Medical Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1210M22861; K12HD068322 (NIH)
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Cystic Fibrosis
Keywords: Biomarkers
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, BALF and Sputum.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CF Infant Cohort: Infants with CF followed for the first two years of life.
- CF Child/Adult Cohort: CF patients > 8 years of age followed during hospitalization for pulmonary exacerbation and when well for two years.

SUMMARY:
Cystic fibrosis (CF) is the most common autosomal recessive genetic disease in Caucasians. It results in lung disease that affects quality of life and causes early death. Lung damage from CF starts in infancy and continues over time. Lung damage can negatively affect how the lung functions. It would be ideal to measure lung damage in CF patients in three instances: (1) During the first year of life after diagnosis by state newborn screening programs, (2) In children and adults over long periods of time (years), and (3) During times of illness (pulmonary exacerbation), to allow for better treatment and therapy to prevent loss of lung function. The lung is made of elastin, collagen and cartilage. When the lung is damaged by CF, these components break down into pieces that can be measured in urine, sputum and blood. These products may represent markers of lung injury. We believe that the levels of these markers will be increased over time in CF patients and even higher in patients who are sick with lung symptoms. The goal of my research is to measure the amount of lung breakdown products in urine, sputum and blood in infants, children and adults with CF during times when well and also during times of illness. I also hope to use new technologies involving the study of proteins and metabolites in samples like sputum, urine and blood to help provide new information regarding CF lung disease. These studies will help us to better treat CF lung disease.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study of two CF populations (and appropriate control populations):

Infants with CF Diagnosed by Newborn Screen: The purpose of this prospective cohort study is to measure concentrations of biomarkers of lung injury in urine, blood and bronchial alveolar lavage fluid (BALF) from CF infants. We plan to characterize these concentrations during the first two years of life with the goal of determining if their profiles alone or in combination are potentially useful biomarkers of early lung disease in CF.

Each CF infant enrolled has blood, urine and BALF samples, along with an oropharyngeal swab (throat culture) in conjunction with infant lung function testing at approximately 6 months of age and again at one year. Our CF Center performs infant Pulmonary Function Tests (PFT's), throat culture and a blood draw as part of routine care at 6 months and at one year of age, so the bronchoscopy and urine collection are obtained for research purposes only. Urine is collected quarterly during routine outpatient clinic visits to the CF Center (4 samples total/year for two years) which is also for research purposes only. During the second year of the study, urine, blood and throat swab sample collection plus lung function testing continue as per year one. In the event of a hospitalization for pulmonary exacerbation, blood and urine samples are obtained at three time points during hospitalization and BALF samples are obtained via bronchoscopy upon admission. An oropharyngeal culture is also obtained upon admission. Subsequent hospitalizations for pulmonary exacerbation are recorded with the same samples collected as described above. In the event of an outpatient exacerbation requiring antibiotic therapy, the patient will be asked to provide a urine sample at the onset of exacerbation. Normal CF treatment or care is not altered in any way by participation in this study.

We collect urine only from age-matched healthy infants as a control group for comparison.

Subjects with CF ≥ 8 Years of Age: The purpose of this prospective cohort study is to measure concentrations of biomarkers of lung injury in urine, blood and sputum from CF patients. This is an observational study that does not involve a specific treatment or intervention. We plan to characterize these concentrations during two years of both clinically stable time points as well during hospitalizations and outpatient treatments for pulmonary exacerbations. The study goal is determining if these profiles alone or in combination are potentially useful biomarkers of early lung disease in CF.

All study participants (CF Exacerbation Group and CF Non-Exacerbation Group) are asked to provide urine, blood and sputum samples, as well as pulmonary function tests, during their regularly scheduled quarterly CF Clinic visits over the study period. Quarterly lung function testing is standard of care for all CF patients. For those patients in the CF Exacerbation group, subjects are asked to provide three urine, blood and sputum samples as well as three sets of pulmonary function before during and after an inpatient hospitalization for a pulmonary exacerbation. We incorporate PFT's, and labs done as part of their hospital admission whenever possible, to avoid duplicate testing. All hospitalized patients will receive their routine, standard-of-care therapies including airway clearance, nutritional support, IV antibiotics and other pulmonary medications. Treatment or care is not be altered in any way by participation in this study. If a patient in the CF Non-Exacerbation Group experiences a pulmonary exacerbation during the study period, samples will be obtained as described for the CF Exacerbation Group.

For a control group comparison we collect sputum and urine only from volunteers > 8 years of age who do not have CF.

ELIGIBILITY:
Infant Study Inclusion Criteria

* Age < 6 months
* Cystic Fibrosis Diagnosed by Newborn Screen

Exclusion:

Age over 6months

Child Study Inclusion Criteria

* FEV1 < 35% predicted A
* Use of IV antibiotics for a pulmonary exacerbation or respiratory symptoms 12 months prior to enrollment.
* Hospitalization for a pulmonary exacerbation 12 months prior to enrollment.
* Use of oral antibiotic for respiratory symptoms 28 days prior to enrollment.
* Any changes in medical regimen for treatment of CF (e.g. no addition of or elimination of therapies such as hypertonic saline, inhaled corticosteroids or mucolytic therapy) within 28 days of enrollment visit.

Exclusion Criteria:

* FEV1 < 35% predicted A
* Use of IV antibiotics for a pulmonary exacerbation or respiratory symptoms 12 months prior to enrollment.
* Hospitalization for a pulmonary exacerbation 12 months prior to enrollment.
* Use of oral antibiotic for respiratory symptoms 28 days prior to enrollment.
* Any changes in medical regimen for treatment of CF (e.g. no addition of or elimination of therapies such as hypertonic saline, inhaled corticosteroids or mucolytic therapy) within 28 days of enrollment visit.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants with Cystic Fibrosis Diagnosed by Newborn Screen.
  Subjects with Cystic Fibrosis => 8 Years of Age.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Biomarkes of Lung Injury | Two Years
  Desmosine,Clara Cell Protein(CC10) and cathepsin B concentration in biological specimens.

SECONDARY OUTCOMES:
Pulmonary Function | Two Years
  Forced expiratory volume (time) (FEV1) and FEV0.5 decline over two years.
Pulmonary Exacerbations | Two years
  The number of CF pulmonary exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Laguna, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States